CLINICAL TRIAL: NCT05515432
Title: Investigation of Pharmacokinetics, Safety and Tolerability of a Single Oral Dose of BAY 3283142 in Participants With Renal Impairment Compared to an Age, Gender and Weight Matched Control Group in an Open-label Study Design
Brief Title: A Study to Learn How the Study Treatment BAY3283142 Taken as Single Dose by Mouth Moves Into, Through, and Out of the Body, How Safe it is, and How it Affects the Body in Participants With Reduced Kidney Function Compared to Participants With Normal Kidney Function of Similar Age, Gender, and Weight
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21593; 2022-000858-28 (EudraCT Number)
Record Dates: First submitted 2022-07-28; First posted 2022-08-25 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease; Renal Impairment; Healthy Volunteers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mildly impaired renal funtion: eGFR (mL/min/1.73 m^2) ≥60 - <90 (Experimental): Participants with renal impairment
  Interventions: Drug: Single oral dose of BAY3283142 IR (immediate release) tablet
- Moderately impaired renal funtion: eGFR (mL/min/1.73 m^2) ≥30 - <60 (Experimental): Participants with renal impairment
  Interventions: Drug: Single oral dose of BAY3283142 IR (immediate release) tablet
- Severely impaired renal funtion: eGFR (mL/min/1.73 m^2) <30 (Experimental): Participants with renal impairment
  Interventions: Drug: Single oral dose of BAY3283142 IR (immediate release) tablet
- ESRD (end stage renal disease) on dialysis (Experimental): Participants with renal impairment
  Interventions: Drug: Single oral dose of BAY3283142 IR (immediate release) tablet
- Normal renal function (control group): eGFR (mL/min/1.73 m^2) ≥90 (Experimental): Age-, weight-, and gender-matched participants with normal renal function as control group
  Interventions: Drug: Single oral dose of BAY3283142 IR (immediate release) tablet

INTERVENTIONS:
Drug: Single oral dose of BAY3283142 IR (immediate release) tablet — Single oral dose of BAY3283142 in participants with renal impairment compared to an age, gender and weight matched control group in an open-label study design

SUMMARY:
Researchers are looking for a better way to treat people who have chronic kidney disease (CKD).

The kidneys filter extra water and waste out of the blood and make urine. CKD is a long-term, progressive, decrease in the kidneys' ability to filter the blood properly. High blood pressure makes it more likely that the CKD gets worse.

The study treatment BAY3283142 is under development for treating CKD. It activates a protein called soluble guanylate cyclase (sGC) that generates cGMP - a molecule that relaxes blood vessels and is thought to have beneficial effects in CKD.

The participants do not benefit from this study. However, the study will provide information on how to use BAY3283142 in subsequent studies in people with CKD.

In previous studies, BAY3283142 was studied in participants with normal kidney function. As kidneys play a role in removal of drugs from the body, the degree of kidney function could influence the amount of BAY3283142 in the blood. Higher amounts may occur in people with reduced kidney function.

Therefore, the main purpose of this study is to learn how the study treatment BAY3283142 moves into, through, and out of the body in participants with mild to severe reduction of kidney function compared to matched participants with normal kidney function.

To answer this, the researchers will compare:

* the (average) total level of BAY3283142 in the blood (also called AUC).
* the (average) highest level of BAY3283142 in the blood (also called cmax) between the different groups. Participants will be in one of four groups based on how much their kidney function is reduced (mild, moderate, severe, end stage kidney disease) or in the control group.

All participants will take a single dose of BAY3283142 as tablet by mouth. Each participant will be in the study for approximately 4 weeks including an in-house stay of 6 days (with 5 overnight stays). In addition, a screening visit to the study site before the in-house stay is planned.

During the study, the study team will:

* check vital signs
* do physical examinations
* take blood and urine samples
* examine heart health using an electrocardiogram (ECG)
* ask the participants questions about how they are feeling and what adverse events they are having

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 82 years of age inclusive, at the time of signing the informed consent.
* Normal kidney function or at different stages of renal impairment (mild to severe renal impairment, ESRD with hemodialysis or hemodiafiltration).
* Race: White (Note: Clinical Data Interchange Standards Consortium [CDISC] definition of White: Denotes a person with European, Middle Eastern, or North African ancestral origin who identifies, or is identified, as White [FDA]).
* Body mass index (BMI) within the range 18.0 and 35.0 kg/m^2 (both inclusive).
* Body weight equal or above 55 kg.
* Male or female participants; women have to be of non-childbearing potential as defined in Section 10.4.1 (e.g., postmenopausal for at least 1 year, women with bilateral salpingectomy, women with bilateral ovariectomy, and women with hysterectomy).
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Men must agree to use a condom in sexual intercourse with female partner of childbearing potential and not to act as sperm donor for 10 days after dosing.
* eGFR <90 mL/min/1.73 m^2 alculated by the CKD-EPI formula (eGFR must be repeated if screening period >10 days before dosing) 21 to 2 days prior to dosing and patients with ESRD on hemodialysis or hemodiafiltration.
* Stable renal function (e.g., a serum creatinine value determined at least 3 months before the screening visit should not vary by more than 25% from the serum creatinine value determined at the screening visit).
* eGFR ≥90 mL/min/1.73 m^2 calculated by the CKD-EPI formula (eGFR must be repeated if screening period >10 days before dosing) 21 to 2 days prior to dosing.
* Needs to be within the required matching age, gender, and body weight range.

Exclusion Criteria:

* Women of childbearing potential, pregnant or lactating women.
* Medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator.
* Known or suspected liver disorders (including Morbus Gilbert/Meulengracht) and bile secretion/flow (cholestasis).
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations).
* Known severe allergies (e.g., allergies to more than 3 allergens, allergies affecting the lower respiratory tract - allergic asthma, allergies requiring therapy with corticosteroids), urticaria, or significant non-allergic drug reactions.
* Relevant acute diseases within the last 4 weeks prior to intake of study intervention.
* Febrile illness within 2 weeks before intake of study intervention.
* Known tendency for vasovagal reactions (e.g., after venipuncture) or clinically relevant history of syncope.
* History of gastrointestinal surgery, with the exception of appendectomy unless it had been performed within the previous 12 months before screening.
* Acute diarrhea or constipation within 14 days before intake of study intervention.
* Diagnosed malignancy within the past 5 years with exception of completely resected basal cell cancer of the skin (excision >6 months before screening).
* Planned intervention or surgery during the study which might impact the study objectives.
* History of clinically relevant bleeding within the past 3 months.
* Thrombotic disorder.
* Use of systemic or topical medicines or substances which oppose the study objectives
* Regular use of therapeutic or recreational drugs, e.g., carnitine products, anabolics, high dose vitamins (except for indicated medications for renally impaired).
* Use of any herbal products or St. John's Wort within the last 14 days before intake of study intervention.
* Excluded therapies (e.g., physiotherapy, acupuncture, etc.) within 1 week before intake of study intervention.
* Change in chronic medications less than 2 weeks prior to dosing.
* Participation in another clinical study during the preceding 3 months for multiple dose studies and 1 month for single dose studies (last visit of participant to previous study to first treatment of new study).
* Exclusion periods from other studies or simultaneous participation in other clinical studies.
* Previous treatment during this study (allowing previously treated participants to be re-included into the study may lead to bias).
* Clinically relevant findings in the physical examination.
* Positive results for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibodies (anti-HCV) (and with a positive polymerase chain reaction [PCR] result or increased liver transaminases or other signs of liver disease), HIV antibodies 1+2/HIV p24 antigen (HIV-1/2 combi test).
* Positive urine/mouth swab drug screening indicating drug abuse.
* Positive alcohol breath test.
* Special diets preventing the participants from eating the standard meals during the study.
* Physical exercise within 96 h before admission the study site.
* Regular daily consumption of more than 1 L of methylxanthine-containing food or beverages.
* Consumption of methylxanthine-containing beverages or food (e.g., coffee, tea, cola drinks, and chocolate) within 48 h before intake of study intervention.
* Smoking more than 10 cigarettes per day.
* Regular daily consumption of more than 500 mL (male participants) or 250 mL (female participants) of usual beer or the equivalent quantity of approximately 20 g (male participants) or 10 g (female participants) of alcohol in another form.
* Intake of foods or beverages containing alcohol within 96 h before intake of study intervention.
* Donation of more than 100 mL of whole blood or plasma within 4 weeks or 500 mL whole blood within 3 months before intake of study intervention.
* Plasmapheresis within 3 months prior to study intervention.
* Suspicion of drug or alcohol abuse.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
AUC of BAY3283142 | up to 0 - 96 hours post-dose
  AUC(0-tlast) will be used as main parameters if AUC cannot be reliably determined in all participants
AUCu of BAY3283142 | up to 0 - 96 hours post-dose
  AUC(0-tlast)u will be used as main parameters if AUC cannot be reliably determined in all participants
Cmax of BAY3283142 | up to 0 - 96 hours post-dose
Cmax,u of BAY3283142 | up to 0 - 96 hours post-dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) after intake of BAY3283142 | up to 7 days post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com